CLINICAL TRIAL: NCT03738605
Title: Vaginal Laser Therapy for the Management of Genitourinary Syndrome of Menopause of Breast Cancer Survivors: Double-blind Randomized Placebo-controlled Trial
Brief Title: Vaginal Laser Therapy in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Themos Grigoriadis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 767/29-09-2017
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Genitourinary Syndrome of Menopause; Vaginal Atrophy; Breast Cancer; Dyspareunia
MeSH Terms: conditions — Breast Neoplasms; Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Experimental): Microablative Fractional CO2 Laser Therapy (The parameters that will be used are the following: 1) Power: 30 ή 40 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter from 1-3 depending on the treatment status, 5) D-pulse mode.)
  Interventions: Device: Microablative Fractional CO2 Laser Therapy
- Placebo (Placebo Comparator): Placebo therapy (The parameters that will be used are the following: 1) Power: 0.5 watts, 2) Dwell time:1000μs, 3) Spacing 1000 μm, 4) Depth: SmartStak parameter 1, 5) Smart-pulse mode.
  Interventions: Device: Microablative Fractional CO2 Laser Therapy

INTERVENTIONS:
Device: Microablative Fractional CO2 Laser Therapy — 5 laser therapies intravaginally administered will be applied at monthly intervals.
  Other Names: SmartXide2 V2LR, Monalisa Touch, DEKA, Florence, Italy

SUMMARY:
This study evaluates the efficacy of vaginal CO2 laser therapy in breast cancer survivors with symptoms of Genitourinary Syndrome of Menopause. Half of participants will receive active laser therapy, while the other half placebo therapy.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer history
* dyspareunia
* dryness

Exclusion Criteria:

* Active genital infection (i.e herpes, vaginitis)
* Prolapse stage >=2
* Underlying pathologies that could interfere with the protocol compliance

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
10-centimeter Visual Analogue Scale assessing intensity of dyspareunia and dryness | Change from baseline at 1 month post-treatment
  It is a straight line with 2 endpoints "0" and "10". Zero defines "no dyspareunia at all" and "no dryness at all" , while 10 "dyspareunia as bad as it could be" and "dryness as bad as it could be". Participants will draw a line at or between the 2 end points. The distance between zero and drawn line will define the intensity of dyspareunia and dryness

SECONDARY OUTCOMES:
3 days voiding diary | Change from baseline at 1 month post-treatment
  Assesses frequency of urination, amount of urine, presence of urgency and/or urinary incontinence and amount of fluid intake
Day-to Day Impact of vaginal aging questionnaire (DIVA) | Change from baseline at 1 month post-treatment
  It includes 4 domains: activities of daily living (5 items), sexual functioning (5 items), emotional well-being (4 items), self-concept and body image (5-items). Each item of each domain could receive values from 0 to 4. Mean scores are calculated on each of the domain scales. Higher scores indicate greater symptom impact
Patients Global Impression of Improvement | At 1-month post-treatment
  It is a single item questionnaire assessing the impression of participants following the intervention
10-centimeter Visual Analogue Scale assessing intensity of itching, burning and dysuria | Change from baseline at 1 month post-treatment
  It is a straight line with 2 endpoints "0" and "10". Zero defines "no symptom (itching, burning and dysuria) at all" , while 10 "symptom (itching, burning and dysuria) as bad as it could be". Participants will draw a line at or between the 2 end points. The distance between zero and drawn line will define the intensity of itching, burning and dysuria
King's Health Questionnaire (KHQ) | Change from baseline at 1 month post-treatment
  It has 3 sections: 1) general health and overall health related to urinary symptoms with 2 questions, 2) incontinence impact, role limitations, physical limitations, social limitations, personal limitations, emotions, sleep and energy, and severity coping measures with 19 questions and 3) bother or impact of urinary symptoms with 11 questions. Scores of each domain of the 2 sections range from 0 to 100. Scores of the third section range from 0 to 3. Higher scores indicate higher impact of urinary incontinence.
Female Sexual Function Index | Change from baseline at 1 month post-treatment
  It is a questionnaire defining women's sexual function. It includes 6 domains: desire, arousal, orgasm, lubrication, satisfaction and pain. The answer of each Question in each domain are multiplied by a certain factor. Total score is calculated by summing the scores of the all domains with a minimum value of 2 and a maximum of 36. The highest the total score the better is the sexual functioning. Total score above 26.55 defines normal sexual function
Vaginal Maturation Value | 6 months
  It is calculated by defining the percentage of superficial, intermediate and parabasal epithelial cells on the vaginal pap smear, following the formula (1x%superficial)+(0.5x%intermediate)+(0x%parabasal). It may receive values from 0 to 100%.It is considered to be an indicator of the estrogenic stimulation, whereas values of 0-49%, 50-64% and 65-100% indicate absent/low, moderate and high estrogenic effect on the vaginal epithelium, respectively.
Vaginal Health Index Score | 6 months
  It evaluates vaginal elasticity, fluid volume, ph of vaginal fluid, epithelial integrity and moisture. Each one of these may receive scores from 1 to 5. Total score is calculated by summing the 5 scores ranging from 5 to 25. Higher scores indicate better vaginal status.
International Consultation on Incontinence Questionnaire Short Form | 6 months
  it is a questionnaire with 4 questions assessing the amount of leakage, frequency and type of urinary incontinence. Total score is calculated by summing the 3 out of the 4 questions. Higher scores indicate worst urinary incontinence
Modified Sexual Quality of Life Questionnaire-Male | 6 months
  It includes 12 questions assessing the quality of life and sexual satisfaction of the male partner. Each answer may receive values from 1 to 5. The higher the scores the better subjective evaluation of sexual quality of life
Urogenital Distress Inventory 6 | 6 months
  It is a condition specific questionnaire containing 6 questions. The answers of questions assesses the presence of symptoms and the degree of bother on a 4-point scale ("not at all", "a little bit", "moderately" and "greatly" applying to 0, 1, 2 and 3, respectively). Total score is calculated by summing the score of each question. The higher the total score the highest is the symptom bother
Epithelial thickness | 6 months
  Biopsies will be obtained from the lateral vaginal wall. Epithelial thickness (in μ) will be measured by a vertical line between basal layer cells and superficial layers.
Number of blood vessels | 6 months
  Biopsies will be obtained from the lateral vaginal wall. Computerized determination of blood vessels number will be performed
Size of blood vessels | 6 months
  Biopsies will be obtained from the lateral vaginal wall. Computerized determination of the blood vessels size will be performed
Collagen | 6 months
  Biopsies will be obtained from the lateral vaginal wall. Determination of collagen types using immunohistochemistry and microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Athanasiou, Associate Proffesor, Study Director — National and Kapodistrian University of Athens, Greece
Locations (1):
- Urogynecological Unit of Alexandra Hospital, Athens, Greece